CLINICAL TRIAL: NCT05081167
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of REL-1017 Monotherapy for Major Depressive Disorder
Brief Title: A Study to Assess the Efficacy and Safety of REL-1017 as Monotherapy for Major Depressive Disorder (MDD)
Acronym: Reliance III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Relmada Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REL-1017-303
Expanded Access: NCT06009003 (Temporarily not available)
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: REL-1017
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REL-1017 (Experimental): A 75 mg REL-1017 loading dose (three 25 mg REL-1017 tablets) will be administered on Day-1 of the 28-day treatment period. From Day-2 to Day-28, participants will take 25 mg REL-1017.
  Interventions: Drug: REL-1017
- Placebo (Placebo Comparator): Three tablets of matching placebo will be administered on Day-1 of the 28-day treatment period. From Day-2 to Day-28, participants will take 1 placebo tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REL-1017 — REL-1017 tablet
  Other Names: esmethadone
  Arms: REL-1017
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
This is an outpatient, 2-arm, Phase 3, multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of REL-1017 once daily (QD) as a monotherapy for Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 65 years, inclusive.
* Diagnosed with Major Depressive Disorder (MDD) based on Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, DSM-5 (SCID-5) for MDD.
* Current major depressive episode.

Exclusion Criteria:

* Any current and primary psychiatric disorder other than Major Depressive Disorder.
* Severe alcohol or substance use disorder.
* History of bipolar I and II disorder, psychosis, and/or mania.
* Acute or chronic condition that, in the Investigator's opinion, would limit the subject's ability to complete or participate in this clinical study.
* Prior participation in a ketamine, esketamine, dextromethorphan or any other NMDAR- antagonist study, or received esketamine at any time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pappagallo, MD, Study Director — Relmada Therapeutics
Locations (9):
- United States (9):
  - Relmada Site, Maitland, Florida
  - Relmada Site, Miami, Florida
  - Relmada Site, Miami Springs, Florida
  - Relmada Site, Orlando, Florida
  - Relmada Site, Palm Bay, Florida
  - Relmada Site, Chicago, Illinois
  - Relmada Site, Boston, Massachusetts
  - Relmada Site, Watertown, Massachusetts
  - Relmada Site, Austin, Texas

REFERENCES:
- See also: Study Homepage — http://reliancestudies.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | REL-1017 | Placebo
Started | 116 | 116
Completed | 108 | 102
Not Completed | 8 | 14

BASELINE CHARACTERISTICS:
Groups:
- REL-1017 25 mg: A 75 mg REL-1017 loading dose (three 25 mg REL-1017 tablets) will be administered on Day-1 of the 28-day treatment period. From Day-2 to Day-28, participants will take 25 mg REL-1017.
  REL-1017: REL-1017 tablet
- Total: Total of all reporting groups
Arm/Group | REL-1017 25 mg | Placebo | Total
Number analyzed (Participants) | 116 | 116 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (13.0) | 38.7 (12.9) | 37.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 71 | 154
  Male | 33 | 45 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 36 | 82
  Not Hispanic or Latino | 68 | 78 | 146
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 23 | 43
  White | 81 | 84 | 165
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in the MADRS10 Total Score From Baseline to Day 28
Description: Therapeutic efficacy of REL-1017 as monotherapy versus placebo in the Montgomery-Asberg Depression Rating Scale (MADRS10).
  A higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60 with scores above 34 indicating severe depression.
  A negative change from baseline indicates improvement.
Time Frame: Day 28
Population: Full Analysis Set: defined as all subjects who received at least one dose of study medication and were assessed for the primary efficacy endpoint at both Baseline and Day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REL-1017 25 mg | Placebo
Number analyzed (Participants) | 105 | 100
score on a scale | -14.8 (12.4) | -13.9 (10.8)

2. Secondary Outcome: MADRS10 Remission Rate (Total Score ≤10) at Day 28
Description: Therapeutic remission rate with REL-1017 as adjunctive treatment versus placebo in the Montgomery-Asberg Depression Rating Scale (MADRS10). Remission is defined as MADRS10 Total Score ≤10 at Day 28. A higher percentage of remission indicates a higher percentage of subjects with MADRS10 Total Score ≤10 at Day 28.
Time Frame: Day 28
Population: Full Analysis Set: defined as all subjects who received at least one dose of study medication and had the Baseline assessment of the primary efficacy endpoint performed
Measure: Number (95% Confidence Interval); unit: percentage of participants in remission
Arm/Group | REL-1017 25 mg | Placebo
Number analyzed (Participants) | 116 | 116
percentage of participants in remission | 21.6 [15.0 to 29.9] | 16.4 [10.7 to 24.2]

3. Secondary Outcome: MADRS10 Response Rate (Improvement ≥50% Compared With Total Baseline Score) at Day 28
Description: Therapeutic response to REL-1017 as adjunctive treatment versus placebo in the Montgomery-Asberg Depression Rating Scale (MADRS10). Response rate is defined as an improvement ≥50% compared with total Baseline MADRS10 score
Time Frame: Day 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | REL-1017 25 mg | Placebo
Number analyzed (Participants) | 116 | 116
percentage of responders | 38.8 [30.4 to 47.9] | 34.5 [26.5 to 43.5]

ADVERSE EVENTS:
Time Frame: TEAE that starts or worsens at any time after initiation of study drug collected up to 14 days post treatment (Day 42).
Description: A Treatment Emergent Adverse Event (TEAE) is defined as an Adverse Event (AE) that starts or worsens at any time after initiation of study drug collected up to 14 days post treatment (Day 42) as collected in the Safety Analysis Set.
Arm/Group | REL-1017 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/116
Other Adverse Events (participants affected / at risk) | 39/116 | 33/116
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REL-1017 25 mg (N=116) | Placebo (N=116)
Headache (Nervous system disorders) | 13 (20) | 11 (11)
Nausea (Gastrointestinal disorders) | 11 (12) | 6 (6)
Dizziness (Nervous system disorders) | 10 (11) | 5 (7)
COVID-19 (Infections and infestations) | 11 (11) | 3 (3)
Fatigue (General disorders) | 6 (6) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 6 (7) | 3 (3)
Upper respirator tract infection (Infections and infestations) | 2 (2) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT05081167/Prot_SAP_000.pdf